CLINICAL TRIAL: NCT01284452
Title: Efficacy of Moderate Dose Hydrocortisone in Treatment of Severe Sepsis and Septic Shock Patients With Acute Lung Injury/Acute Respiratory Distress Syndrome: A Randomized Controlled Trial
Brief Title: Efficacy of Hydrocortisone in Treatment of Severe Sepsis/Septic Shock Patients With Acute Lung Injury/Acute Respiratory Distress Syndrome (ARDS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Surat Tongyoo, MD, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Si630/2010
Record Dates: First submitted 2011-01-18; First posted 2011-01-27 (Estimated); Last update posted 2015-04-20 (Estimated); Status verified 2015-04

CONDITIONS: Septic Shock; Severe Sepsis; Acute Lung Injury; Acute Respiratory Distress Syndrome
Keywords: Septic shock; Severe sepsis; Acute lung injury; Acute respiratory distress syndrome; ARDS
MeSH Terms: conditions — Shock, Septic; Sepsis; Acute Lung Injury; Respiratory Distress Syndrome | interventions — Hydrocortisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Normal saline 50 ml intravenous every 6 hours for 7 days
  Interventions: Drug: Placebo
- Hydrocortisone (Active Comparator): Hydrocortisone 50 mg intravenous every 6 hours for 7 days
  Interventions: Drug: Hydrocortisone

INTERVENTIONS:
Drug: Placebo — Normal saline 50 ml intravenous every 6 hours for 7 days
  Arms: Placebo
Drug: Hydrocortisone — Hydrocortisone 50 mg intravenous every 6 hours for 7 days
  Arms: Hydrocortisone

SUMMARY:
Severe sepsis/septic shock is a serious condition associated with high mortality rate. Hydrocortisone has been recommended as a useful treatment to decrease mortality in hemodynamically unstable septic shock patients, not response to fluid and moderate dose of vasopressor. During the progression of severe sepsis/septic shock, multi-organ dysfunction can develop. Acute lung injury (ALI) and its more severe form, acute respiratory syndrome (ARDS) is one of the common organ dysfunction associated with septic shock. Information from a meta-analysis suggested that moderate dose of hydrocortisone may improve the ARDS patients' outcome. Whether hydrocortisone can effectively prevent disease progression and death in severe sepsis/septic shock patients who complicated with ALI/ARDS has not been proven.

DETAILED DESCRIPTION:
Severe sepsis/septic shock is a serious condition associated with high mortality rate. The pathophysiology of the disease involves the complex interaction between host's immunity and the microorganisms toxin. The release of immune complex and cascade of inflammatory cytokines are responsible for multiorgan dysfunction, especially the cardiovascular system. Hydrocortisone has been recommended as a useful treatment to decrease mortality in hemodynamically unstable septic shock patients, not response to fluid and moderate dose of vasopressor. Both anti-inflammation and supplementation of relatively adrenal insufficiency are the main hypothesis of the benefit of hydrocortisone. During the progression of severe sepsis/septic shock, multi-organ dysfunction can develop. Acute lung injury (ALI) and its more severe form, acute respiratory syndrome (ARDS) is one of the common organ dysfunction associated with septic shock. Although there is controversy about timing and favorable patients'characteristic, the information from a meta-analysis suggested that moderate dose of hydrocortisone may improve the ARDS patients' outcome. Whether hydrocortisone can effectively prevent disease progression and death in severe sepsis/septic shock patients who complicated with ALI/ARDS has not been proven.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Diagnosis of severe sepsis or septic shock according to the American College of Chest Physicians/Society of Critical Care Medicine Consensus Conference 1992
* Diagnosis of acute lung injury or acute respiratory distress syndrome according to the American-European Consensus Conference on ARDS 1994
* Onset of organ dysfunction within 12 hours before enrollment

Exclusion Criteria:

* Indicated for receive corticosteroid
* Congestive heart failure
* Contra-indication for hydrocortisone: For example: allergy to hydrocortisone
* Pregnancy
* Not agree to sign the consent form

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2010-12; Primary Completion 2014-12 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
All cause mortality | 28 days
  Death from any cause at 28 days after diagnosis of severe sepsis/septic shock

SECONDARY OUTCOMES:
Ventilator free day | 28 day
  Day of alive within 28 days without mechanical ventilator support.
Vasopressor free day | 28 days
  Days of alive within 28 days without any doses of vasopressors including dopamine, norepinephrine, adrenaline or dobutamine.
Rate of renal replacement therapy | 28 days
  Proportion of the patients who received renal replacement therapy within 28 days after diagnosis of severe sepsis or septic shock.
Organ support free days | 28 days
  Days of alive without ventilator, renal replacement therapy and vasopressors within 28 days after diagnosis of severe sepsis or septic shock.

CONTACTS AND LOCATIONS:
Overall Officials: Surat Tongyoo, MD, Principal Investigator — Department of Medicine, Faculty of Medicine Siriraj Hospital, Mahidol University
Locations (1):
- Department of Medicine, Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok, Bangkok, Thailand

REFERENCES:
- [Derived] Tongyoo S, Permpikul C, Mongkolpun W, Vattanavanit V, Udompanturak S, Kocak M, Meduri GU. Hydrocortisone treatment in early sepsis-associated acute respiratory distress syndrome: results of a randomized controlled trial. Crit Care. 2016 Oct 15;20(1):329. doi: 10.1186/s13054-016-1511-2. PMID 27741949